CLINICAL TRIAL: NCT00975845
Title: A Prospective, Double-Blind Evaluation of the Effects of BioCleanse Tibialis Tendon Allograft and Donor Age on Clinical Outcomes of ACL Reconstruction
Brief Title: BioCleanse Tibialis Tendon Anterior Cruciate Ligament (ACL) Study
Status: Completed | Type: Observational
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: BCTib 2008
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: ACL; Anterior Cruciate Ligament; Torn tendon; ACL Repair; ACL reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BioCleanse Tibialis Tendon Allograft: Tibialis Tendon allograft from donor 18-65 years old
  Interventions: Other: BioCleanse Tibialis tendon

INTERVENTIONS:
Other: BioCleanse Tibialis tendon — Outcomes of anterior cruciate replacement will be evaluated

SUMMARY:
To compare the outcome of Anterior Cruciate Ligament (ACL) reconstruction performed using the tibialis allograft to historical outcomes of ACL reconstruction patients and to establish if any correlation exists between the age of the graft donor and the clinical outcomes.

DETAILED DESCRIPTION:
This is a single-arm, single site, pilot study in patients with a ruptured ACL. A total of fifty (50) subjects will be enrolled in this trial. All patients will have been scheduled to undergo ACL reconstruction and will receive a BioCleanse Tibialis allograft as part of the normal standard of care practiced by the treating surgeon. Follow up is for 2 years.

However, there is no assignment of graft, specific to donor age, to the patients. All treatment will follow standard of care and this study assumes that there will be a normal distribution of graft donor ages, from 18 to 65 years of age.

Patient outcomes will be compared between the 2 groups of tendon donor ages. Neither the surgeon nor the patient will be aware of the age of the graft donor, per typical standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Study subjects will be limited to those subjects undergoing allograft anterior cruciate ligament reconstruction surgery
2. Meniscal injuries may be included
3. Isolated, unilateral anterior cruciate ligament injury.
4. All subjects will have a minimum age of eighteen (18) years and a maximum of sixty (60) years.
5. Both male and non-pregnant female subjects will be included.
6. To facilitate follow-up, study subjects will be limited to the local geographic area of the study site and be willing to use the rehabilitation facility and physical therapy schedule assigned by the surgeon.
7. All subjects must be able to read, write, and comprehend instructions and guidelines in English and understand (and sign as an acknowledgment of their understanding) an informed consent declaration.

Exclusion Criteria:

1. No chondral defects
2. Failure to comply with or meet all of the inclusion criteria listed above.
3. Autograft anterior cruciate ligament surgery on either knee.
4. Anterior cruciate ligament injury on contra-lateral leg at any time
5. Multi-ligament reconstruction
6. Inability to comply with all requirements of this investigation, as well as follow the instructions of the physician.
7. Significant systemic disease or conditions which impact overall health or well being or which necessitate chronic medication use.
8. Revision anterior cruciate ligament surgery to either knee at anytime
9. Exhibiting signs of moderate to severe degenerative joint disease in addition to requiring anterior cruciate ligament surgery.
10. Concomitant injuries to the knee or lower extremities requiring treatment, per surgeon's discretion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who have had reconstruction of the anterior cruciate ligament and have received a BioCleanse Tibialis allograft for ACL reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Objective International Knee Documentation Committee (IKDC) Exam | pre-op, 2 months, 4 months, 6 months, 12 months, 24 months
  The International Knee Documentation Committee (IKDC) is a knee-specific patient-reported outcome measure. This is an indexed score form 0-100, with 0 being the worst possible status and 100 indicating no dysfunction, disability or pain.

SECONDARY OUTCOMES:
Subjective quality of life scores | pre-op, 2 months, 4 months, 6 months, 12 months, and 24 months
  The SF36 measures the quality life as reported by the paritricpantm, and is an indexed score form 0 - 100. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Carter, MD, Principal Investigator — Foundation for Orthopedic Research and Education
Locations (1):
- The Orthopedic Clinic, Assoc, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No